CLINICAL TRIAL: NCT03806504
Title: Prospective Randomized Trial of Impact of High PEEP Application Following Pulmonary Endarterectomy on Outcome
Brief Title: High PEEP Application Following Pulmonary Thromboendarterectomy; Does it Have Any Impact on Outcome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, mustafa emre gürcü, anesthesia and reanimation specialist, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018/6/62
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Reperfusion Injury After Pulmonary Thromboendarterektomy
Keywords: Chronic thromboembolic pulmonary hypertension; PEEP; reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: prospective, randomized
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high PEEP (Active Comparator): 35 cm/H2O PEEP, 2-3 ml/kg tidal volume,45 seconds, after cardiopulmonary bypass
  Interventions: Other: PEEP
- control group (Active Comparator): 6 cm/H2O PEEP, 6-8 ml/kg tidal volume, continues, after cardiopulmonary bypass
  Interventions: Other: control group

INTERVENTIONS:
Other: PEEP — performing 35 cm/H2O PEEP and 2-3 ml/kg tidal volume
  Arms: high PEEP
Other: control group — performing 6 cm/H2O PEEP and 6-8 ml/kg tidal volume
  Arms: control group

SUMMARY:
Investigation of the effect of intraoperative lung protection high PEEP maneuver on ischemic reperfusion injury in patients undergoing pulmonary endarterectomy.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a rare disease characterized by progression of thromboembolism obstructing pulmonary arteries as an organized tissue. Pulmonary thromboendarterectomy (PTE) is a treatment option for chronic thromboembolic pulmonary disease. However, PTE is associated with specific postoperative complications, such as pulmonary edema and right ventricular failure due to reperfusion injury, with a significant mortality rate of 7% to 24%. Some strategies have been proposed to reduce lung injury after PTE, such as rectification maneuvers and high PEEP. The aim of this study was to investigate the effect of intraoperative lung protection high PEEP maneuver in patients undergoing pulmonary endarterectomy for ischemic reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective PTE operation due to CTEPH,
* 20-70 years old

Exclusion Criteria:

* Patients with chronic inflammatory disease,
* liver and renal failure,
* heart failure (<EF: 40%),
* intraoperative bronchial hemorrhage,
* patients undergoing postoperative revision.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
free oxygen radicals levels | 48 hours
  Superoxide dismutase (SOD) activity will be measured by modification of the method of Sun et al. and Protein carbonyl groups will be determined by volume modification according to Reznick and Packer method.

SECONDARY OUTCOMES:
postoperatif outcome - Duration of stay in the intensive care unit and hospital stay | 10 day
  Duration of stay in the intensive care unit and hospital stay after pte operation

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa EMRE Gurcu, Istanbul, Turkey (Türkiye)